CLINICAL TRIAL: NCT06542211
Title: Observation on the Efficacy of Improving Ankle Dorsiflexion Limitation in Patients With Plantar Fasciitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2023360
Record Dates: First submitted 2024-08-04; First posted 2024-08-07 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-05

CONDITIONS: Plantar Fasciitis
Keywords: ankle dorisflexion; plantar fasciitis
MeSH Terms: conditions — Fasciitis, Plantar

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plantar Fasciitis Test Group (Experimental): The experimental group received intervention and rehabilitation training directly for the limited ankle dorsiflexion function, which mainly included subtalar joint loosening (increasing the joint activity space), plantar flexor muscle group relaxation (releasing the tension of antagonist muscles), ankle dorsiflexor muscle strengthening (enhancing the strength of agonist muscles), and integrated exercises (integrating ankle dorsiflexion function into gait training).
  Interventions: Behavioral: Intervention plan for improving ankle dorsiflexion limitation group (experimental group)
- Plantar fasciitis conventional rehabilitation group (Active Comparator): Conventional rehabilitation for plantar fasciitis mainly focuses on relaxing the plantar fascia, gastrocnemius and plantar flexor muscles and strengthening the small muscle groups of the plantar foot.
  Interventions: Behavioral: Plantar fasciitis routine rehabilitation group

INTERVENTIONS:
Behavioral: Intervention plan for improving ankle dorsiflexion limitation group (experimental group) — The experimental group received intervention and rehabilitation training directly for the limited ankle dorsiflexion function, which mainly included subtalar joint loosening (increasing the joint activity space), plantar flexor muscle group relaxation (releasing the tension of antagonist muscles), ankle dorsiflexor muscle strengthening (enhancing the strength of agonist muscles), and integrated exercises (integrating ankle dorsiflexion function into gait training).
  Arms: Plantar Fasciitis Test Group
Behavioral: Plantar fasciitis routine rehabilitation group — The experimental group received intervention and rehabilitation training directly for the limited ankle dorsiflexion function, which mainly included subtalar joint loosening (increasing the joint activity space), plantar flexor muscle group relaxation (releasing the tension of antagonist muscles), ankle dorsiflexor muscle strengthening (enhancing the strength of agonist muscles), and integrated exercises (integrating ankle dorsiflexion function into gait training).
  Arms: Plantar fasciitis conventional rehabilitation group

SUMMARY:
This study aims to design a randomized controlled trial to treat plantar fasciitis by combining conventional rehabilitation with the improvement of ankle dorsiflexion function, and to explore its clinical efficacy by combining various evaluation indicators.

Compared with conventional plantar fasciitis, ankle dorsiflexion function rehabilitation training focuses more on the improvement of patients' foot and ankle function. Conventional PF rehabilitation training focuses on loosening the plantar fascia and gastrocnemius muscle, which can restore the elasticity of the plantar fascia and promote pain relief, but has limited improvement in ankle dorsiflexion function, resulting in patients' daily life such as walking, squatting, and going upstairs. Ankle dorsiflexion function rehabilitation training is an intervention directly targeting the function of the foot and ankle joint. By restoring the ankle dorsiflexion function of patients, it helps patients correct the force line in daily life movements, reduce the probability of sports injury risk, and improve sports performance and daily life satisfaction.

Conventional rehabilitation for plantar fasciitis mainly focuses on relaxing the plantar fascia, gastrocnemius muscle, and plantar flexor muscle strength and strengthening the small muscle group exercises of the plantar foot.

The experimental group directly intervened and conducted rehabilitation training for the limited ankle dorsiflexion function. It mainly includes subtalar joint loosening (increasing joint activity space), plantar flexor muscle group relaxation (releasing antagonist muscle tension), ankle dorsiflexor muscle strengthening (enhancing agonist muscle strength), and integrated exercises (integrating ankle dorsiflexion function into gait training).

This experiment lasted for a total of eight weeks, and patients were required to complete five home rehabilitation training sessions per week.

DETAILED DESCRIPTION:
Plantar fasciitis (PF) is a common musculoskeletal injury characterized by inflammation and degeneration at the origin of the fascia and causing heel pain. The disease affects individuals of different ages and activity levels and is the main cause of plantar pain and ankle dysfunction in patients, accounting for 15% of all foot diseases. A previous study showed that PF is more common in middle-aged and elderly people and those who love sports. One in 10 people has their daily quality of life seriously affected by PF. In clinical work, it was found that there was a large difference in the degree of ankle function of PF patients at the time of consultation. The clinical symptoms of plantar fasciitis are mainly heel pain when landing in the morning or after a long rest. The symptoms are aggravated after standing or walking for a long time, and sometimes patients will show a pain-reducing gait. The diagnosis is mainly based on the patient's symptoms and signs. There are often local tenderness points when palpating along the plantar fascia and the medial tubercle of the calcaneus. The patient's ankle dorsiflexion range of motion may be limited. Ultrasound examination shows increased thickness of the plantar fascia. The patient may also show bone spurs growing into the fascia on X-rays . The cause of plantar fasciitis is still unclear. Its risk factors include age, obesity, foot deformity, limited ankle dorsiflexion, decreased foot proprioception, long-term weight-bearing and walking activities . These factors are interrelated and interact with each other, and the abnormal biomechanical mechanism of the foot is the key to the internal connection between these factors . Poor foot-ankle force line and biomechanics will increase abnormal stress on the plantar fascia during joint movement, leading to micro-tears of the fascia, and then thickening and tightening of the plantar fascia, resulting in inflammation. At present, the intervention treatment methods for plantar fasciitis are divided into two categories: surgery and conservative treatment. Most patients are treated with conservative treatment, which mainly includes insole adjustment, physical therapy and weight loss. Physical therapy programs generally include stretching the plantar fascia and calf muscles, muscle strength training, taping, the use of orthotics and night splints, etc.. Currently, the short-term effect is acceptable, but the long-term effect is poor, and it is easy to relapse, which affects the overall motor function and sports performance.

People have higher and higher requirements for health. In addition to paying attention to local pain relief, patients with plantar fasciitis also have higher demands for improving sports performance. Conventional physical therapy methods can effectively relieve the temporary pain of patients with plantar fasciitis, but the recovery of patients' motor function is still poor. Only relieving short-term pain symptoms can no longer fully meet people's daily life and sports needs. For the long-term rehabilitation of plantar fasciitis, the correction of poor foot biomechanics and the improvement of foot and ankle function are the key to preventing and improving physical function and improving sports performance. Ankle dorsiflexion dysfunction will reduce various sports performances and increase the compensation of other joint functions in the body, thereby increasing the risk and probability of sports injuries. Relevant studies have shown that limited ankle dorsiflexion is one of the causes of plantar fasciitis. A study showed that 211 out of 254 patients had limited ankle dorsiflexion . Individuals with insufficient ankle dorsiflexion during walking may roll their feet forward by dropping the talus and flattening the medial longitudinal arch. The flattening of the arch may stretch the plantar fascia, which may lead to inflammation of the plantar fascia over time . However, the current treatment methods for plantar fasciitis have failed to systematically improve the limited ankle dorsiflexion function of patients, and limited ankle joint function may directly affect the long-term treatment effect of plantar fasciitis.

In summary, since the correction of poor foot force line and the recovery of ankle dorsiflexion function play an important role in the long-term treatment effect of plantar fasciitis, this study aims to design a randomized controlled trial to treat plantar fasciitis in combination with conventional rehabilitation and improvement of limited ankle dorsiflexion function, and to explore its clinical efficacy in combination with various evaluation indicators.

ELIGIBILITY:
Inclusion Criteria:

1. Age range: 30-60 years old; disease course > 3 months; pain cannot be relieved by conservative treatment such as rest, oral nonsteroidal drugs, and physical therapy; VAS score is less than 6 points.
2. According to the clinical practice guidelines of the International Classification of Functioning, Disability and Health: Heel Pain/Plantar Fasciitis: 2014 Revision [16], patients meet the clinical diagnostic criteria for PF, mainly including pain on the medial side of the plantar, heel pain caused by recent weight-bearing activities, pain on palpation of the proximal attachment of the plantar fascia, and positive Windlass test;
3. Supine straight knee ankle dorsiflexion angle <10°; lunge knee flexion <40° [50, 51]; left and right foot dorsiflexion difference does not exceed 1°.
4. BMI between 18.5-23.9 (Chinese standard)

Exclusion Criteria:

- (1) Those who have received local injections of steroids in the past 3 months; (2) Those with other foot, ankle and lower leg diseases: history of surgery, fracture, trauma, plantar skin ulcers, rheumatism or rheumatoid arthritis, etc.; (3) Those with serious medical diseases: such as blood diseases, coagulopathy, severe cardiovascular and cerebrovascular dysfunction, tumor diseases, etc.

(4) Those with peripheral neuropathy (idiopathic, diabetic, nutritional); L5/S1 neural foramen impingement or lumbar spinal stenosis (5) Congenital structural flat feet, equinus deformity or other foot and ankle joint diseases

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2025-03-02 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
Vicon 3D gait test | 40min
  The subjects wore sports shorts, fully exposing the waist and the area below the mid-thigh. After the reflective markers were fixed, the subjects first familiarized themselves with the requirements and process of collecting movements according to the test procedures. The subjects stood in the center of the test room, with their feet shoulder-width apart and their upper limbs naturally placed on both sides of the body. They kept the subtalar joint in a neutral position and conducted three static tests to collect static data for defining the coordinate system of the bone segments. Afterwards, the subjects performed walking and jogging tests at the speed they felt most comfortable. The interval between the two tests was based on the patient not feeling tired. 5 valid data were collected for each action, and the average value of the 5 tests was used for analysis.
Plantar fascia thickness measurement | 20min
  The Japanese KONICA MINOLTA musculoskeletal ultrasound was used for testing, with a probe frequency of 3 to 18 Hz. Experienced clinicians were selected to perform the measurements. The patients were placed in a prone position with their ankle joints in a neutral position. The calcaneus and plantar fascia junction were measured. The doctor measured the plantar fascia thickness on the affected side of the patient, and the average value of three ultrasound measurement images was selected each time.
Ankle dorsiflexion angle measurement | 10min
  Ankle dorsiflexion angle in supine straight knee position and in lunge with bent knee position

SECONDARY OUTCOMES:
Ankle and hindfoot function rating scale | 10min
  American Orthopedic Foot Ankle Society (AOFAS) Ankle and Hindfoot Function Rating Scale: The scale is commonly used for rehabilitation assessment of foot pain and function, including 9 items: pain, function and autonomous activity, support, maximum walking distance (block), ground walking, abnormal gait, front and back activity (flexion and extension), hindfoot activity (inversion-extension), ankle-hindfoot stability (front and back and inversion-extension), foot force line. The total score of the scale is 100 points, no conversion is required, just add them up directly.
  The grading standard is: excellent, 90-100 points; good, 75-89 points; acceptable, 50-74 points; poor, <50 points.
Visual Analogue Scale for Pain | 20min
  The VAS pain visual analogue scale is a simple and clear method for pain statistics. It is one of the most commonly used scales for clinical pain statistics and is used to evaluate and monitor the degree of heel pain in patients before and after treatment. Draw a 10cm long horizontal line on the paper, with the starting end of the line at "0", representing no pain; the end of the line at "10", representing severe pain; the middle part of the line represents different degrees of pain; ask the patient to self-assess the heel pain when taking the first step in the morning and draw the corresponding position on the horizontal line.
Plantar pressure test | 20min
  The subjects walked barefoot on a footscan® pressure plate (RSscan, 2×0.4 m, 16,384 sensors) at a self-selected speed. The pressure plate was placed in the middle of a 30-m runway. Before the test, the subjects warmed up and became familiar with the barefoot walking procedure, and then took the test at a self-selected appropriate speed. If the heel did not touch the ground first during a test or the subject's walking speed differed from the average of their normal walking speed by more than 10%, the test was considered invalid and the subject was asked to retest. Five valid test data were collected from each foot for analysis.
  The plantar pressure standardization method proposed by Keijsers et al. [8] was used for analysis: each foot was first scaled and rotated, and then the plantar pressure of each sensor was standardized with the plantar pressure of the whole foot.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No